CLINICAL TRIAL: NCT02001194
Title: A Randomized Trial of Behavioral Economic Interventions to Improve Physical Activities: Team Incentives
Brief Title: Way to Be Active I (Teams)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 819101
Record Dates: First submitted 2013-11-27; First posted 2013-12-04 (Estimated); Results first posted 2019-03-05 (Actual); Last update posted 2019-03-05 (Actual); Status verified 2019-02

CONDITIONS: Sedentary Employees
Keywords: Sedentary; Behavioral Economic Intervention; Team Studies; Financial Incentives; Workplace Wellness; Team Incentives
MeSH Terms: conditions — Sedentary Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Control (No Intervention): Participants receive either an email or text message daily (based on the participant's preference) stating whether the participant achieved the 7000 step goal during the previous day. Each participant will also be notified as to how many of their teammates reached the goal the previous day. Control Arm will receive no financial incentive.
- Individual (Experimental): Participants receive either an email or text message daily (based on the participant's preference) stating whether the participant achieved the 7000 step goal during the previous day. Each participant will also be notified as to how many of their teammates reached the goal the previous day. Every day one team from the arm will be chosen at random as the winning team. Each participant on the winning team receives $50 if that participant met the step goal during the prior day.
  Interventions: Behavioral: Individual Incentives
- Team (Experimental): Participants receive either an email or text message daily (based on the participant's preference) stating whether the participant achieved the 7000 step goal during the previous day. Each participant will also be notified as to how many of their teammates reached the goal the previous day. Every day one team from the arm will be chosen at random as the winning team. Each participant on the winning team receives $50 only if all four team members met the step goal during the prior day.
  Interventions: Behavioral: Team Incentives
- Individual Plus Team (Experimental): Participants receive either an email or text message daily (based on the participant's preference) stating whether the participant achieved the 7000 step goal during the previous day. Each participant will also be notified as to how many of their teammates reached the goal the previous day. Every day one team from the arm will be chosen at random as the winning team. Each participant on the winning team receives $20 if the participant met the step goal during the prior day the participants met their own goal. Each participant will also receive an additional $10 for every one of the other three team members that also met the goal.
  Interventions: Behavioral: Individual plus Team Incentives

INTERVENTIONS:
Behavioral: Individual Incentives
  Arms: Individual
Behavioral: Team Incentives
  Arms: Team
Behavioral: Individual plus Team Incentives
  Arms: Individual Plus Team

SUMMARY:
Employers are increasingly looking for opportunities to motivate sedentary employees to become more physically active. Workplace walking programs have had mixed success and typically show most improvement among participants that are already fairly active at a baseline. The goal of this study is to determine whether a financial incentive program can motivate sedentary employees to increase the number of steps they walk per day to meet a minimum threshold.

Our primary outcome measure is the proportion of days a minimum activity of 7000 steps or more is achieved. We will assess outcomes each week for 3 months using incentives followed by 3 months of follow-up without incentives. Secondary outcomes will include the average steps walked per day.

ELIGIBILITY:
Inclusion Criteria:

* 1. We will use a minimum age of 18 to ensure all individuals are legally able to consent.
* 2. Participant will need an iPhone or Android smartphone to be able to use the Moves App for tracking steps

Exclusion Criteria:

* Conditions that would make participation infeasible: 1a. Inability to consent 1b. Illiteracy and/or inability to speak, read, and write English 1c. Participation in another research study 2. Conditions that would make participation unsafe: 2a. Current treatment for drug or alcohol use 2b. Consumption of at least 5 alcoholic drinks per day 2c. Myocardial infarction or stroke within the past 6 months 2d. Current addiction to prescription medicines or street drugs 2e. Serious psychiatric diagnoses (e.g., severe major depressive disorder, bipolar disorder, schizophrenia) 2f. Pregnant or currently breastfeeding 2g. Metastatic cancer 2h. Unstable medical conditions that would likely prevent the participant from completing the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Actual)
Dates: Start 2014-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

REFERENCES:
- [Derived] Patel MS, Asch DA, Rosin R, Small DS, Bellamy SL, Eberbach K, Walters KJ, Haff N, Lee SM, Wesby L, Hoffer K, Shuttleworth D, Taylor DH, Hilbert V, Zhu J, Yang L, Wang X, Volpp KG. Individual Versus Team-Based Financial Incentives to Increase Physical Activity: A Randomized, Controlled Trial. J Gen Intern Med. 2016 Jul;31(7):746-54. doi: 10.1007/s11606-016-3627-0. Epub 2016 Mar 14. PMID 26976287

RESULTS

PARTICIPANT FLOW:
Groups:
- Individual: Participants receive either an email or text message daily (based on the participant's preference) stating whether the participant achieved the 7000 step goal during the previous day. Each participant will also be notified as to how many of their teammates reached the goal the previous day. Every day one team from the arm will be chosen at random as the winning team. Each participant on the winning team receives $50 if that participant met the step goal during the prior day.
  Individual Incentives
- Team: Participants receive either an email or text message daily (based on the participant's preference) stating whether the participant achieved the 7000 step goal during the previous day. Each participant will also be notified as to how many of their teammates reached the goal the previous day. Every day one team from the arm will be chosen at random as the winning team. Each participant on the winning team receives $50 only if all four team members met the step goal during the prior day.
  Team Incentives
- Individual Plus Team: Participants receive either an email or text message daily (based on the participant's preference) stating whether the participant achieved the 7000 step goal during the previous day. Each participant will also be notified as to how many of their teammates reached the goal the previous day. Every day one team from the arm will be chosen at random as the winning team. Each participant on the winning team receives $20 if the participant met the step goal during the prior day the participants met their own goal. Each participant will also receive an additional $10 for every one of the other three team members that also met the goal.
  Individual plus Team Incentives
Period: Intervention Period (13 Weeks)
Arm/Group | Control | Individual | Team | Individual Plus Team
Started | 68 (17 teams) | 80 (20 teams) | 76 (19 teams) | 80 (20 teams)
Completed | 67 (16 teams) | 80 (20 teams) | 74 (19 teams) | 78 (20 teams)
Not Completed | 1 | 0 | 2 | 2
Not completed — No longer interested | 1 | 0 | 2 | 2
Period: Follow-Up Period (13 Weeks)
Arm/Group | Control | Individual | Team | Individual Plus Team
Started | 67 | 80 | 74 | 78
Completed | 64 | 78 | 73 | 78
Not Completed | 3 | 2 | 1 | 0
Not completed — No longer interested | 3 | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Individual | Team | Individual Plus Team | Total
Number analyzed (Participants) | 68 | 80 | 76 | 80 | 304
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (10.0) | 39.3 (10.2) | 38.7 (10.2) | 41.2 (10.8) | 40.6 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 62 | 65 | 57 | 235
  Male | 17 | 18 | 11 | 23 | 69
Marital Status [Count of Participants; unit: Participants]
  Single | 28 | 43 | 33 | 26 | 130
  Married | 35 | 29 | 32 | 41 | 137
  Other | 5 | 8 | 11 | 13 | 37
Education [Count of Participants; unit: Participants]
  Less than college | 2 | 7 | 6 | 7 | 22
  Some college | 20 | 23 | 26 | 21 | 90
  College graduate | 45 | 50 | 44 | 52 | 191
  Unknown | 1 | 0 | 0 | 0 | 1
Annual Household Income [Count of Participants; unit: Participants]
  Less than $50,000 | 9 | 21 | 13 | 11 | 54
  $50,000 to $100,000 | 24 | 34 | 38 | 34 | 130
  Greater than $100,000 | 27 | 18 | 21 | 30 | 96
  Unknown | 8 | 7 | 4 | 5 | 24
iPhone smartphone [Count of Participants; unit: Participants] | 40 | 47 | 43 | 55 | 185
Race/Ethnicity [Count of Participants; unit: Participants]
  White non-Hispanic | 38 | 30 | 43 | 50 | 161
  African American non-Hispanic | 22 | 37 | 23 | 19 | 101
  Other non-Hispanic | 3 | 9 | 6 | 8 | 26
  Hispanic | 5 | 4 | 3 | 3 | 15
  Missing | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Days a Minimum Activity of 7000 Steps or More is Achieved
Description: Our primary outcome measure is the proportion of days a minimum activity of 7000 steps or more is achieved. We will assess outcomes for 3 months (13 weeks) with the interventions and 3 months (13 weeks) without intervention during the follow-up period. We will use all available data and treat missing as true missing data points. Secondary outcomes will include the average steps walked per day.
Time Frame: End of study- 6 months of after enrollment
Measure: Mean (95% Confidence Interval); unit: Proportion of participant-days
Arm/Group | Control | Individual | Team | Individual Plus Team
Number analyzed (Participants) | 68 | 80 | 76 | 80
Proportion of participant-days
  Intervention Period | 0.176 [0.101 to 0.250] | 0.254 [0.185 to 0.322] | 0.173 [0.103 to 0.243] | 0.350 [0.281 to 0.419]
  Follow Up Period | 0.142 [0.068 to 0.215] | 0.187 [0.120 to 0.255] | 0.152 [0.082 to 0.221] | 0.235 [0.167 to 0.302]

2. Secondary Outcome: Average Number of Steps Per Day During Intervention
Description: Secondary outcomes include average number of steps per day during intervention period and the follow-up period.
Time Frame: End of study- 6 months after enrollment
Measure: Mean (95% Confidence Interval); unit: steps per day
Arm/Group | Control | Individual | Team | Individual Plus Team
Number analyzed (Participants) | 68 | 80 | 76 | 80
steps per day
  Intervention Period (3 months with incentives) | 3929.1 [3170.5 to 4687.7] | 4516.4 [3817.1 to 5215.8] | 3929.6 [3212.1 to 4647.4] | 5280.3 [4580.9 to 5979.7]
  Follow Up Period (3 months without incentives) | 3619.1 [2827.3 to 4410.8] | 3957.8 [3227.8 to 4687.7] | 3713.1 [2964.1 to 4462.0] | 4616.0 [3886.1 to 5346.0]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected during the intervention (weeks 1-13) and the follow-up phase of the study (weeks 14-26).
Arm/Group | Control | Individual | Team | Individual Plus Team
All-Cause Mortality (participants affected / at risk) | 0/68 | 0/80 | 0/76 | 0/80
Serious Adverse Events (participants affected / at risk) | 0/68 | 0/80 | 0/76 | 0/80
Other Adverse Events (participants affected / at risk) | 0/68 | 0/80 | 0/76 | 0/80

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No